CLINICAL TRIAL: NCT03564964
Title: An Intermediate-Size, Expanded Access to SUVN-502 for the Treatment of Subjects With Alzheimer's Disease Who Have Completed the CTP2S1502HT6 Study
Brief Title: Expanded Access to Provide SUVN-502 for the Treatment of Subjects With Alzheimer's Disease
Acronym: SUVN-502
Status: No longer available | Type: Expanded Access
Sponsor: Suven Life Sciences Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: EAP1502HT6
Record Dates: First submitted 2018-05-28; First posted 2018-06-21 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Alzheimer Disease; Dementia; Cognition Disorders
Keywords: SUVN-502; Expanded Access
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognition Disorders | interventions — 1-((2-bromophenyl)sulfonyl)-5-methoxy-3-((4-methyl-1-piperazinyl)methyl)-1H-indole dimesylate monohydrate

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: SUVN-502 — Tablet

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide access to SUVN-502 for the treatment of Alzheimer's Disease. Investigator as well as the subject/caregiver must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the patient's medical history and program eligibility criteria.

Subjects will not be evaluated for efficacy and safety during the expanded access.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed the 30 week treatment period of study CTP2S1502HT6 as planned and wish to continue treatment with SUVN-502.
* Subject (or subject's legally acceptable representative) and caregiver must sign the Informed Consent Form (ICF) to participate in the study.

Exclusion Criteria:

* Has participated or is participating in any other clinical (investigational) study after completion of CTP2S1502HT6 study.
* Is treated or likely to require treatment during the study with any medication prohibited by this expanded access program.

Ages: 50 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult